CLINICAL TRIAL: NCT05313230
Title: Safety and Efficacy of Intermittent Renal Replacement Therapy Using CITRASATE in Critically-ill Patients: A Retrospective Series
Brief Title: Safety and Efficacy of Intermittent Renal Replacement Therapy Using CITRASATE in Critically-ill Patients
Acronym: CITRA-SAFE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0739
Record Dates: First submitted 2022-01-06; First posted 2022-04-06 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Acute Kidney Injury; Chronic Kidney Infection
Keywords: Renal Replacement Therapy; CITRASATE
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CITRASAFE: Patient underwent CITRASATE dialysis session
  Interventions: Other: CITRASATE SLED

INTERVENTIONS:
Other: CITRASATE SLED — Applying of CITRASATE SLED

SUMMARY:
Renal Replacement Therapy (RRT) needs an extracorporeal circulation to conduct blood to the dialysis membrane and driving back to the patient. This extracorporeal circulation induces inevitably a risk of coagulation activation and premature clotting of the circuit. Heparin is thereby commonly used to prevent such thrombosis but exposed patient to risk of hemorrhage. This risk of hemorrhage may be important in ICU population, particularly in severe trauma patients.

The calcium is an important determinant of coagulation cascade. The use of specific citrate enriched dialysate without calcium (CITRASATE®) allows to suddenly lower the calcium concentration in extracorporeal plasma, leading to a regional ineffectiveness of clotting and limited heparin needs. This low calcium plasmatic concentration into the extracorporeal circulation has however to be normalized to not generate a systemic hypocalcemia. In our ICU, a local calcium substitution protocol based on dialysate flow is used in clinical practice.

Commonly used in our unit, there is a lack data to evaluate the CITRASATE dialysate in a critical population.

The aim goal of our study will be to assess safety and efficacy of intermittent renal replacement therapy using CITRASATE® in critically-ill patients.

DETAILED DESCRIPTION:
This is a retrospective descriptive study. The included patients will be those who had a Sustained Low Efficiency Dialysis using CITRASATE® dialysate in CHU Lapeyronie in Montpellier, France between 01/01/2019 and 31/12/2021 Using PMSI code, we estimate that 61 patients could be enrolled in this period and each patient could be almost 6 dialysis session. We estimate we could analyzed 300 to 350 sessions. This sample must be confirmed by the opening of medical records.

A data collection will be focused on the RRT parameters, clinical complications until ICU discharge and outcome, extracted from medical records.

The main endpoint will be to determine the prevalence of ionized calcium troubles (hypocalcemia <0,8 mmol/L or Hypercalcemia >1,4 mmol/L) per and post dialysis using CITRASATE® with our restitution protocol, and their therapeutic consequences.

The secondary endpoints will be to describe the efficacy of CITRASATE® with our restitution protocol during RRT meant by an optimal dialysis dose and the absence of premature clotting of the circuit.

ELIGIBILITY:
Inclusion criteria:

* Age ≥18 years
* Patient underwent a RRT in the DAR Lapeyronie (CHU Montpellier) between the 01/01/2019 and the 31/12/2021

Exclusion criteria:

* Patient underwent RRT without CITRASATE® protocol
* Lack of data
* Ethical limitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient underwent a RRT in the DAR Lapeyronie (CHU Montpellier) between the 01/01/2019 and the 31/12/2021
Sampling Method: Non-Probability Sample
Enrollment: 61 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
change of blood ionized calcium level disorders | baseline, per dialysis session
  Retrospective assessment of the prevalence of ionized calcium troubles (hypocalcemia <0,8 mmol/L or Hypercalcemia >1,4 mmol/L) per and post-dialysis using CITRASATE® with our restitution protocol, and their therapeutic consequences.
change of blood ionized calcium level disorders | Day 1 (post dialysis session)
  Retrospective assessment of the prevalence of ionized calcium troubles (hypocalcemia <0,8 mmol/L or Hypercalcemia >1,4 mmol/L) per and post-dialysis using CITRASATE® with our restitution protocol, and their therapeutic consequences.

SECONDARY OUTCOMES:
Description of therapeutic consequences required | day 1
  therapeutic consequences required in order to treat the ionized calcium troubles
Description of Clotting event | day 1
  the efficacy of CITRASATE® with our restitution protocol during RRT absence
Description of Dialysis dose | day 1
  the efficacy of CITRASATE® with our restitution protocol during RRT (optimal dialysis dose)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan CHARBIT, MD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, Montepllier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC